CLINICAL TRIAL: NCT03276156
Title: Apatinib in Combination With S-1 as Second-Line Treatment in Patients With Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Apatinib in Combination With S-1 as Second-Line Treatment in Patients With Advanced Gastric Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ahead-G001
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib plus S-1 (Experimental): Apatinib (425/500/675/750mg,qd,p.o.) concomitantly with S-1 (80mg to 120 mg, qd,days1-14, q3w, p.o.)
  Interventions: Drug: Apatinib plus S-1

INTERVENTIONS:
Drug: Apatinib plus S-1 — Drug:Apatinib (425 mg/d) + S-1 (80mg to 120 mg);Drug:Apatinib (500 mg/d) + S-1 (80mg to 120 mg);Drug:Apatinib (675mg/d) + S-1 (80mg to 120 mg);Drug:Apatinib (750 mg/d) + S-1 (80mg to 120 mg);

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD)and safety of Apatinib combined with S-1 as Second-line therapy for patients with advanced gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed consent prior to any specific research procedure.
2. Adult patients, aged ≥18 years;
3. Imaging test confirmed the progression after first-line treatment of advanced gastric adenocarcinoma or Gastroesophageal Junction Adenocarcinoma.

   * S-1 was not used in the first-line treatment
   * If patient relapse in 6 months after adjuvant chemotherapy or neoadjuvant chemotherapy, the adjuvant chemotherapy or neoadjuvant chemotherapy was regarded as the first-line treatment.
4. Adjuvant chemotherapy or neoadjuvant chemotherapy was allowed if the first-line treatment started beyond 6 months after the end of previous treatment.
5. During the research ,patient should be willing and be able to follow the process treatment ,follow up and tests.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.
7. Survival expectation ≥ 16 weeks from the planned first dosing .
8. During the 28 days prior to the first dosing, hematological, biochemical and Organ Functions:HB ≥ 9.0 g/dL, ANC ≥ 1.5×109/L,WBC>3×109/L， PLT ≥ 100×109/L, BIL < 1.5×ULN, ALT or AST < 2.5×ULN (or < 5×ULN in patients with liver metastases), Serum Cr ≤ 1.5×ULN;
9. Lesions ,measurable and/or unmeasurable,at least one,can be assessed by imaging during the baseline and follow-up measurement.

   * Localized mass in gastric or Gastroesophageal Junction belongs to unmeasurable Lesions.
10. Women, those postmenopausal or of child-bearing age, but the pregnancy test results (serum or urine) within 28 days before treatment is negative, and the results should be confirmed in day 1 of the treatment.

    * Postmenopausal women are defined as :woman's menstrual periods have ceased for 1 year or longer after exogenous hormone therapy;
    * Women, aged>50years,serum LH and FSH level show a postmenopause;
    * Woman has radiation induced ovarian failure,and gone without a period for over 12 consecutive months;
    * Woman has chemotherapy-induced menopause and gone without a period for over 12 consecutive months;
    * sterilization operation( hysterectomy or bilateral oophorectomy)

Exclusion Criteria:

1. Has participated in another clinical trial in progress.
2. Has received more than one chemotherapy regimens after disease progression(except for those who has receiced adjuvant chemotherapy or neoadjuvant chemotherapy 6 months or longer)
3. Previous therapy with S-1
4. Has received VEGFR inhibitor, such as Sorafenib,Sunitinib .
5. Has another primary tumor,but adequately treated non-melanoma skin cancer , effectively treated carcinoma in situ of cervix and other well handled cancer over 5 years were not covered.
6. Has difficulty in swallowing
7. Has taken experimental drugs within 14 days before randomly assign.( For different drug characteristics, the interval can be longer)
8. History of any chemotherapy, radiotherapy,the last administration should finish within 3 weeks prior to trial first drug administration( For different drug characteristics, the interval can be longer). If steady dose of diphosphate or denosumab is necessary for the treatment of bone metastases,the administration should start 3-4weeks prior to the study .
9. Patients with poor-controlled arterial hypertension (systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mm Hg) despite standard medical management; Coronary heart disease greater than Class I, arrhythmia greater than Class I (including QT interval prolongation, for man > 450 ms, for woman > 470 ms), and cardiac dysfunction greater than Class I;
10. Has persistent toxicity (exclude alopecia )of previous treatment ,CTCAE>1.
11. Has intestinal obstruction or upper gastrointestinal hemorrhage(CTCAE 3 or 4) within 4 weeks prior to randomly assign.
12. Abnormal coagulation function (INR > 1.5×ULN, APTT > 1.5×ULN), with tendency of bleed;
13. Has symptom of brain metastases and the tendency out of control,but imaging confirmed is not required.If steady dose of Glucocorticoid is necessary for the treatment,the administration should be started >4weeks prior to the study . Patients with spinal cord compression received definite treatment and the situation had been proven stable in 28days .
14. Has surgery within 2 weeks prior to the study. Eligible patients should recovered from any major surgery.
15. Subjects that are unable to swallow tablets, chronic diarrhea ,or intestinal obstruction;
16. Subjects with a clear tendency of gastrointestinal bleeding;
17. Pregnant or lactating women;
18. Other conditions regimented at investigators' discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-02-23 (Actual); Primary Completion 2018-02-22 (Estimated); Study Completion 2018-02-22 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | Event driven, an expected average of 4 months
Incidence of adverse events | An expected average of 4 months

SECONDARY OUTCOMES:
Overall survival(OS) | An expected average of 12months
Disease control rate(DCR) | An expected average of 4 months
Objective response rate(ORR) | An expected average of 4 months
Quality of life(QoL) | An expected average of 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China